CLINICAL TRIAL: NCT01025726
Title: Improving Safety and Access for Physical Activity
Brief Title: Positive Action for Today's Health
Acronym: PATH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Dawn Wilson, Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Pro00005110; R01DK067615 (NIH)
Record Dates: First submitted 2009-12-01; First posted 2009-12-03 (Estimated); Last update posted 2023-01-19 (Actual); Status verified 2012-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Social Marketing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Full Intervention (Experimental): Police Patrolled Walking Program plus Social Marketing Intervention
  Interventions: Behavioral: Police Patrolled Walking plus Social Marketing
- Walking Only (Experimental): Police Patrolled Walking Only Intervention
  Interventions: Behavioral: Police Patrolled Walking Program Only
- General Health (Active Comparator): General Health Education Intervention
  Interventions: Behavioral: General Health Education

INTERVENTIONS:
Behavioral: Police Patrolled Walking plus Social Marketing — Identify walking route, hire walking leaders and police support, maintain route and monitor stray dogs PLUS grass-roots social marketing campaign to promote walking on the route
  Arms: Full Intervention
Behavioral: Police Patrolled Walking Program Only — Identify walking route, hire walking leaders and police support, maintain route and monitor stray dogs
  Arms: Walking Only
Behavioral: General Health Education — Host community events for chronic disease education
  Arms: General Health

SUMMARY:
Regular moderate and vigorous intensity physical activity (PA) is inversely related with obesity, however, few adults are successful in incorporating sufficient PA into their daily lives. Minority and lower-income adults have among the highest obesity rates and lowest levels of regular PA. Increasing environmental supports for safe and convenient places for PA is an emerging public health strategy for PA interventions. Preliminary data by Wilson (PI) and colleagues has revealed through focus groups that low-income minority adults would like to increase the safe places for PA (areas free from crime, containment of stray dogs, increased police patrol) and access to PA (sidewalks/trails and expand opportunities for PA) in their community. In addition, the results of the investigators' preliminary studies suggest that African Americans had psychosocial barriers to PA that included lack of self-motivation, cultural body image issues, and lack of time due to family obligations. The present proposal is innovative in that it specifically tests the efficacy of an intervention that includes both patrolled-walking and social marketing elements to increase PA in low-income African Americans. Three communities will be randomized to receive one of three programs: a police patrolled-walking program plus social marketing intervention, a police patrolled-walking only intervention, or no walking intervention (general health education only; N=390; 130/group). The 24-month intervention will focus on increasing safety (training community leaders to serve as walking captains, hiring off-duty police officers to patrol the walking program, and containing stray dogs), increasing access for PA (marking a walking route), and will include a tailored social marketing campaign for increasing PA (in one intervention community). The investigators will collect data for PA (7-day accelerometer estimates, 4-week PA history), body composition, blood pressure, psychosocial measures, and perceptions of environmental supports for safety and access for PA at baseline, 6-,12-,18-, and 24-months. The primary hypotheses are that the patrolled-walking plus social marketing intervention will result in greater increases in moderate and vigorous PA as compared to a patrolled walking only intervention or no-intervention by 12-months and that these effects will be maintained at 18-month and 24-month assessments.

ELIGIBILITY:
Inclusion Criteria:

* African American (3 of 4 grandparents are of African Descent)
* Lives in designated census area
* No plans to move in the next two years
* Has no medical condition that would limit participation in moderate intensity exercise including life-threatening illness (e.g., immobile, severely disabled, or bed ridden)
* Available and able to participate in measures and intervention activities over the next 2 years

Exclusion Criteria:

* Extreme Blood Pressure and/or Blood Glucose levels
* Unable to take a brisk, 30-minute walk

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 439 (Actual)
Dates: Start 2007-07; Primary Completion 2011-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Physical Activity (Accelerometer) | 0, 6, 12, 18, 24 months

SECONDARY OUTCOMES:
Blood Pressure | 0, 6, 12, 18, 24 months
Body Mass Index (BMI) | 0, 6, 12, 18, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Dawn K Wilson, PhD, Principal Investigator — University of South Carolina
Locations (3):
- United States (3):
  - Pee Dee CAP Weed & Seed, Florence, South Carolina
  - Ministry of Reconcilliation, Orangeburg, South Carolina
  - M.H. Newton Family Life Enrichment Center, Sumter, South Carolina

REFERENCES:
- [Derived] McDaniel T, Wilson DK, Coulon MS, Sweeney AM, Van Horn ML. Interaction of Neighborhood and Genetic Risk on Waist Circumference in African-American Adults: A Longitudinal Study. Ann Behav Med. 2021 Jul 22;55(8):708-719. doi: 10.1093/abm/kaaa063. PMID 32914830
- [Derived] Abshire DA, Wilson DK, Sweeney AM, Pinto BM. Correlates of Moderate-to-Vigorous Physical Activity and Exercise Motivation in Underserved African American Men. Am J Mens Health. 2019 May-Jun;13(3):1557988319855155. doi: 10.1177/1557988319855155. PMID 31148501
- [Derived] Sweeney AM, Wilson DK, Lee Van Horn M. Longitudinal relationships between self-concept for physical activity and neighborhood social life as predictors of physical activity among older African American adults. Int J Behav Nutr Phys Act. 2017 May 22;14(1):67. doi: 10.1186/s12966-017-0523-x. PMID 28532489
- [Derived] Wilson DK, Van Horn ML, Siceloff ER, Alia KA, St George SM, Lawman HG, Trumpeter NN, Coulon SM, Griffin SF, Wandersman A, Egan B, Colabianchi N, Forthofer M, Gadson B. The Results of the "Positive Action for Today's Health" (PATH) Trial for Increasing Walking and Physical Activity in Underserved African-American Communities. Ann Behav Med. 2015 Jun;49(3):398-410. doi: 10.1007/s12160-014-9664-1. PMID 25385203